CLINICAL TRIAL: NCT04612946
Title: Using Connected Health to Increase Lung Cancer Screening: Single Center Randomized Pilot Trial
Brief Title: Using Connected Health to Increase Lung Cancer Screening
Acronym: CH-LCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 844390
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer
Keywords: telemedicine; behavioral economics; connected health strategies; lung cancer screening; patient outreach
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomized (1:1) intervention or usual care
Who Masked: Outcomes Assessor
Masking Description: Primary analyst and statistician will be blinded to the randomization assignment. The investigators and research coordinators will be unblinded to facilitate coordination with telehealth referral. The analyst will create the randomization assignments on a master list (using Stata) and enter into REDCap using the randomization module (stratified by batch). Assignments will be maintained by the research coordinator on a password protected computer. The blind may be broken in the case of an emergency.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Patients in the intervention arm will be invited to complete a telemedicine LCS counseling visit and asked for permission to be referred (name and phone number) to the LCS navigator at Penn Medicine to schedule a telemedicine visit. Patients will also be given the option to directly contact the LCS navigator.
  Interventions: Behavioral: Referral to Telemedicine LCS Counseling Visit
- Control Arm (Active Comparator): Patients in the usual care arm will be provided with contact information for the Penn LCS Program and encouraged to discuss LCS with their primary care providers.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Referral to Telemedicine LCS Counseling Visit — Patients in the intervention arm will be invited to complete a telemedicine LCS counseling visit, and asked for permission to be referred directly to the LCS navigator to help schedule an appointment. They will also be given the option to directly contact the LCS navigator. Telemedicine counseling visits will be conducted using established clinical procedures for virtual or telephone visits at Penn Medicine. In accordance with reimbursement policies for lung cancer screening, these visits will be conducted by a physician or nurse practitioner within the Lung Cancer Screening Program at Penn Medicine. Counseling visits are covered without co-pay as standalone visits according to USPSTF guidelines and costs will not be covered by the study. LCS is an evidence-based practice and considered standard of care for those who are eligible and desire to be screened. Clinicians retain full control on how to conduct LCS counseling or LDCT in this trial.
  Arms: Intervention Arm
Behavioral: Usual Care — Patients in the usual care arm will be provided with contact information for the Penn LCS Program and encouraged to discuss LCS with their providers.
  Arms: Control Arm

SUMMARY:
This study will consist of two primary aims designed to help advance quality and utilization of lung cancer screening (LCS) within an academic and community-based medical system. The objective of Aim 1 is to pilot test the effect and feasibility of using direct outreach and telemedicine to increase LCS counseling and LDCT uptake among screening-eligible patients. Patients who confirm eligibility and agree to participate will be randomized into two study arms: 1) usual care or 2) telemedicine LCS counseling referral. For Aim 2, each arm will first complete a baseline survey to explore how individual beliefs and knowledge impact screening intention and uptake. Patients in both arms will also receive brief information on lung cancer screening guidelines and be asked to report LCS-related preferences after exposure to the information. All interventions will be administered using a secure, web-based platform.

DETAILED DESCRIPTION:
In 2013, the United States Preventive Services Task Force (USPSTF) provided a Grade "B" recommendation for annual lung cancer screening (LCS) for asymptomatic adults aged 55-80 who are or have been heavy smokers (≥30 pack-years of smoking and quit-date < 15 years ago), and are able to undergo surgery. In 2015, The Centers for Medicare and Medicaid Services (CMS) issued national coverage for LCS requiring that LCS counseling, which must include shared decision-making and tobacco cessation counseling, occur prior to LCS. CMS also provides reimbursement for LCS counseling to further support providers to engage in meaningful, collaborative conversations about LCS with patients. Despite widespread support, uptake and implementation of LCS across the United States has been low (estimated 3-5% screening-eligible population screened). Locally, since the onset of the Penn Medicine LCS Program in 2014, over 3,500 individual patients have received LCS; however, documentation and reimbursement of LCS counseling are limited.

Challenges of implementing LCS include substantial barriers to identifying screening-eligible patients, supporting high-quality decision-making, and remaining uncertainties regarding risks and benefits. For other types of cancer screening, insights from behavioral science have been applied to understand how cognitive biases and beliefs impact screening uptake. Yet for LCS, there is limited evidence on how these beliefs may affect screening behaviors in routine practice. Given the complexities of LCS, in which the benefits do not clearly outweigh the harms, understanding how these biases impact screening can help inform development of intervention strategies that both support informed decision-making and increase uptake among eligible patients. Leveraging an existing EMR-based data warehouse, this study will combine insights from behavioral economics and connected health strategies to pilot test connected health approaches including direct patient outreach and telemedicine visits to improve LCS counseling, and to explore individual-level moderators of LCS screening intention and uptake. The long-term goal is to decrease lung cancer burden by increasing utilization of LCS and providing clinicians and patients with effective strategies to deliver high-quality, patient-centered care. This study will also advance scientific understanding of the mechanisms that drive or hinder health behavior in the context of cancer prevention.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 55-77
2. Had a primary care visit at the healthcare system within the last 24 months
3. No history of lung cancer
4. Heavy smokers (30+ pack year and current smoker or quit within 15 years)
5. Access to phone and internet
6. English-speaking
7. Have an assigned primary care provider at recruiting practices
8. Never received LCS within the healthcare system

Exclusion Criteria:

1. Aged <55 or >77 years
2. Did not have a primary care visit at the healthcare system within the last 24 months
3. History of lung cancer
4. Smoking history of <30 pack years
5. No access to phone and internet
6. Inability to speak English
7. Does not have an assigned primary care provider at recruiting practices
8. History of LCS within the healthcare system

Ages: 55 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Completion of LCS counseling | Initial measurement will occur within 8 weeks of baseline survey
  The primary outcome measure is completion of LCS counseling, defined by completion of a telemedicine visit, in-person counseling visit (CPT G0296), or documentation of counseling in EHR provider notes.

SECONDARY OUTCOMES:
Completion of LDCT scan for LCS | Within 6 months following baseline survey
  The secondary outcome is completion of LDCT scan for LCS as captured in the EHR.

CONTACTS AND LOCATIONS:
Overall Officials: Katharine A Rendle, PhD,MSW,MPH, Principal Investigator — University of Pennsylvania; Anil Vachani, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We do not have any plans to share IPD at this time, but we are open to sharing de-identified data with other researchers as allowed and approved by our institutional review board and following our planned analysis and publications.

REFERENCES:
- [Derived] Rendle KA, Steltz JP, Cohen S, Schapira MM, Wender RC, Bekelman JE, Vachani A. Estimating Pack-Year Eligibility for Lung Cancer Screening Using 2 Yes or No Questions. JAMA Netw Open. 2023 Aug 1;6(8):e2327363. doi: 10.1001/jamanetworkopen.2023.27363. PMID 37548980

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT04612946/Prot_SAP_000.pdf